CLINICAL TRIAL: NCT03595670
Title: Illness Representations in Patients With Bipolar Disorders. What Mecanisms and What Impacts on Adherence and Quality of Life ?
Brief Title: Illness Representations in Patients With Bipolar Disorders
Acronym: RsBiP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-55
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group: • Patients diagnosed bipolar in mania, depression or euthymic phases according DSM-IV critiera by psychiatrist
  standardized questionnaires and interview will be performed
  Interventions: Other: standardized questionnaires; Other: interview

INTERVENTIONS:
Other: standardized questionnaires — standardized questionnaires concerning the perception
Other: interview — Semi-directive interviews will be conducted. The purpose of this approach is to question the meaning of the disease (beliefs, representations), the psycho-social management of the disease, its inscription in the socio-cultural condition of the patients.

SUMMARY:
Bipolar disorder is a serious and chronic illness representing a major health problem with high mortality rates. According to the self-regulation model , patients had some representations of their illness which are cognitive and emotional. Cognitive representations include the set of beliefs built around the illness, its consequences and treatment. Emotional representations are negative emotions generated by the presence of the illness. According to Leventhal et al. (1997), representations are linked to information extracts by patients from society, relatives, experiences. This model has been particularly studied in the context of somatic disorders, but Baines & Wittkowski (2013) shown that it may also be relevant in patients with mental disorders. In bipolar disorders, first results show that illness representations are related to relapses and to medication adherence. That's why, we think that this relevant to improve knowledges of the psychological processes that accompany the experience of bipolar disorders. To assess illness representation, we will use both qualitative and quantitative tools. These results could have direct application to clinical practice in psychosocial interventions.

DETAILED DESCRIPTION:
Bipolar disorder is a serious and chronic illness representing a major health problem with high mortality rates (Colom and Lam, 2005). According to the self-regulation model (Leventhal, Nerenz & Steel, 1986), patients had some representations of their illness which are cognitive and emotional. Cognitive representations include the set of beliefs built around the illness, its consequences and treatment. Emotional representations are negative emotions generated by the presence of the illness. According to Leventhal et al. (1997), representations are linked to information extracts by patients from society, relatives, experiences. This model has been particularly studied in the context of somatic disorders, but Baines & Wittkowski (2013) shown that it may also be relevant in patients with mental disorders. In bipolar disorders, first results show that illness representations are related to relapses (Lobban et al., 2013) and to medication adherence (Averous, Charbonnier, Lagouanelle-Simeoni, Prosperi & Dany, 2018). That's why, we think that this relevant to improve knowledges of the psychological processes that accompany the experience of bipolar disorders. To assess illness representation, we will use both qualitative and quantitative tools. These results could have direct application to clinical practice in psychosocial interventions.

ELIGIBILITY:
Inclusion Criteria:

* Men or women whose is between 18 and 85 years
* Patients diagnosed bipolar in mania, depression or euthymic phases according DSM-IV critiera by psychiatrist
* Taking in charge in the framework of service Psychiatrie Secteur 5 - Hôpitaux Sud - Hôpital Sainte Marguerite de Marseille
* Patients agreeing to participate to study

Exclusion Criteria:

* Minor patients or over 85 years old
* Patients not understanding French
* Patients with neurological or psychiatric disorders prohibiting their comprehension of the study
* Patients deprived of their liberty following a judicial or administrative decision
* Patients supported without their consent
* Patients under legal guardianship
* Patients treated in emergencies
* Patients refusing to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed bipolar in mania, depression or euthymic phases according DSM-IV critiera by psychiatrist
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-11 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Illness perception for schizophrenia (IPQS) | 24 hours
  IPQS in an autoquestionnaire evaluating illness representations according to the self-regulation model.

SECONDARY OUTCOMES:
Illness Perception Questionnaire Bref (IPQ-B) | 24 hours
  IPQ-B evaluate similar dimensions from IPQ-S in only once item.
Qualitative study of illness perceptions | 24 hours
  Measure of illness representations according to the self-regulation model evaluated with a semi-structured interview.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France